CLINICAL TRIAL: NCT01646632
Title: Effects of Exercise on ADL Performance, Physical Fitness, and Care Dependency in Institutionalized Elderly People
Brief Title: Exercise Intervention in Institutionalized Elderly People
Acronym: BENENFIT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hanze University of Applied Sciences Groningen (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Mrs. Elizabeth Weening-Dijksterhuis, researcher, Hanze University of Applied Sciences Groningen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABR NL 24558.042.09
Record Dates: First submitted 2012-07-11; First posted 2012-07-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Fragility; Physical Disability
Keywords: institutionalized ADL fitness care-dependency
MeSH Terms: interventions — Resistance Training; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical exercise intervention (Experimental): Progressive resistance training, balance training, functional training
  Interventions: Behavioral: Physical exercise intervention
- Lifestyle counseling (Placebo Comparator): Recreational sessions
  Interventions: Behavioral: Lifestyle counseling

INTERVENTIONS:
Behavioral: Physical exercise intervention — the experimental intervention included group- based progressive resistance training, balance training, and functional training, two times a week, one hour sessions, lasting 16 weeks.
  Other Names: strength training; muscle training; coordination training
  Arms: Physical exercise intervention
Behavioral: Lifestyle counseling — the control intervention included recreational sessions, including talks, video's, music, board games etc. No physical activity was involved in the control intervention.
  Other Names: leisure time activities without physical activity
  Arms: Lifestyle counseling

SUMMARY:
Questions: Does an evidence-based exercise program increase activities of daily living and physical fitness in institutionalized older adults? Does this program decrease the care dependency of institutionalized older adults? Design: A randomized control trial using group-based exercise was performed in 14 assisted-living facilities for the elderly (>70 years old).

Outcome measures: Outcome measures were performance on ADL, physical fitness, and care dependency measures. The exercise program comprised group-based progressive resistance training, balance training, and functional training. The control intervention comprised social group meetings.

DETAILED DESCRIPTION:
To improve physical fitness, a combined exercise program including progressive resistance training, balance training, and functional training will be used in a sample of institutionalized elderly people. The exercise program has a frequency of 2 times a week and a duration of 16 weeks. The intensity is moderate, measured on a 0-10 scale. The level of intensity is specified as follows: on a 10- point scale, where no movement is 0 and maximal effort of a muscle group is 10, moderate-intensity effort is a 5 or 6, and high- intensity effort is a 7 or 8. There is currently insufficient evidence that a combined exercise program, developed to improve physical fitness, can improve ADL performance and care dependency also.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 and older
* Being able to walk at least 10 meters
* Not cognitive impaired

Exclusion Criteria:

* Dementia
* Severe hart failure
* Progressive neurological diseases

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 164 (Actual)
Dates: Start 2009-10; Primary Completion 2012-12 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
ADL performance in institutionalized elderly people | 16 weeks
  the intervention was either an group -based exercise program (the experimental intervention), or a recreational program (the control intervention), lasting 16 weeks, two times a week, including one hour sessions

SECONDARY OUTCOMES:
Physical fitness in institutionalized older people | 16 weeks
  the intervention was either an group -based exercise program (the experimental intervention), or a recreational program (the control intervention), lasting 16 weeks, two times a week, including one hour sessions
Care dependency in institutionalized older people | 16 weeks
  the intervention was either an group -based exercise program (the experimental intervention), or a recreational program (the control intervention), lasting 16 weeks, two times a week, including one hour sessions

CONTACTS AND LOCATIONS:
Overall Officials: Cees P van der Schans, Prof., PhD, Study Chair — Hanze University Applied Science Groningen The Netherlands
Locations (1):
- Hanze University Applied Sciences, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Background] Weening-Dijksterhuis E, Kamsma YP, van Heuvelen MJ. Psychometric properties of the PAT: an assessment tool for ADL performance of older people living in residential homes. Gerontology. 2011;57(5):405-13. doi: 10.1159/000318151. Epub 2010 Aug 26. PMID 20798482
- [Background] Weening-Dijksterhuis E, de Greef MH, Scherder EJ, Slaets JP, van der Schans CP. Frail institutionalized older persons: A comprehensive review on physical exercise, physical fitness, activities of daily living, and quality-of-life. Am J Phys Med Rehabil. 2011 Feb;90(2):156-68. doi: 10.1097/PHM.0b013e3181f703ef. PMID 20881587